CLINICAL TRIAL: NCT03023488
Title: Effects Of Flexible Ureteroscopy On Renal Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MAR.UAD.002; 09.2016.181 (Other: Clinical Research Ethics Committee of Marmara University)
Record Dates: First submitted 2016-02-11; First posted 2017-01-18 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Circulatory; Change
Keywords: flexible ureteroscopy; blood flow
MeSH Terms: interventions — Lithotripsy, Laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flexible ureteroscopy arm (Experimental): the findings of patients undergoing flexible ureteroscopy + laser lithotripsy for renal stones according to EAU Guidelines Doppler Ultrasound examination has been performed in the pre-operative and post-operative periods
  Interventions: Procedure: flexible ureteroscopy; Device: Doppler Ultrasound examination; Device: laser lithotripsy

INTERVENTIONS:
Procedure: flexible ureteroscopy — Flexible ureteroscopy is an endourological procedure performed for kidney stones. The flexible ureteroscope is a device used to reach the renal cavities through the natural urinary tract in a retrograde fashion. During the operation, irrigation fluid is used to expand the cavities to provide space for movement of the device and also to provide clear vision.
Device: Doppler Ultrasound examination — peak systolic velocities (PSV) and end diastolic velocities (EDV) of the arteries will be measured and then resistive index (RI) and pulsatility index (PI) will be calculated.
Device: laser lithotripsy — The laser fiber extending into the cavities through the working channel of the ureteroscope is used to fragment the stones. Laser energy is generated by the laser machine and transmitted to the stones via the laser fiber.

SUMMARY:
Aim of this study is to investigate the effects of increased intrarenal pressure during flexible ureteroscopy on renal blood flow.

Patients undergoing flexible ureteroscopy (F-URS) and laser lithotripsy for kidney stones according to European Association of Urology (EAU) guidelines on Urolithiasis will be included in the study after having signed an informed consent form. The pre- and post-operative evaluation and management will be performed according to EAU Guidelines on Urolithiasis. Additionally, as a non-invasive test, bilateral renal power Doppler US will be performed to patients pre- and post-operatively. The pre-operative Doppler US will be performed 2 days prior to surgery and the post-operative Doppler US will be performed in the first 24 hours following surgery. The changes on blood flow in renal artery and arcuate artery will be recorded.

DETAILED DESCRIPTION:
Aim of this study is to investigate the effects of increased intrarenal pressure during flexible ureteroscopy on renal blood flow.

Patients undergoing flexible ureteroscopy and laser lithotripsy for kidney stones according to EAU guidelines on Urolithiasis will be included in the study after having signed an informed consent form. The pre- and post-operative evaluation and management will be performed according to EAU Guidelines on Urolithiasis. Additionally, as a non-invasive test, bilateral renal power Doppler US will be performed to patients pre- and post-operatively. The pre-operative Doppler US will be performed 2 days prior to surgery and the post-operative Doppler US will be performed in the first 24 hours following surgery. The changes on blood flow in renal artery and arcuate artery will be recorded.

Flexible ureteroscopy has been a key component of kidney stone management in the last 20 years. Even for stones larger than 2 cm, flexible ureteroscopy can be performed with high success and low complication rates. Ureteral access sheaths are key contributors to flexible ureteroscopy as they provide easy and repeated access to upper urinary tract and decreased intrarenal pressures due to easy flow back of the irrigation solution.

The increased pressures during flexible ureteroscopy have been an important research area in the last years. Due to irrigation solution and irrigational pumping to provide a clearer vision during flexible ureteroscopy, intrarenal pressures rise and after a certain point pyelo-sinusoidal, pyelo-venous and pyelo-lymphatic backflow starts. It has been shown that this backflow starts when pressure rises above 40 cmH2O (centimeters-water / unit of pressure measurement). Schwalb et al. demonstrated in their study that in kidneys subject to high intrarenal pressure, denudation and flattening of the caliceal urothelium, submucosal edema and congestion are observed. Due to these deleterious effects on urothelium, renal extravasation and bacterial translocation can occur and complications may arise.

Renal Doppler US, due to its non-invasive nature, has been widely used to measure localized blood flow in the kidneys, to evaluate hemodynamic parameters in acute kidney injury. Intrarenal backflow and its consequences such as submucosal edema and congestion may decrease blood flow especially around the calyces subject to high pressures and this situation may result in acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients between ages 18-65
* Patients undergoing flexible ureteroscopy + laser lithotripsy according to EAU Guidelines on Urolithiasis

Exclusion Criteria:

* Pregnant patients
* Patients with already-diagnosed urological malignancies
* Patients ineligible for flexible ureteroscopy due to concomitant co-morbidities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarik Emre Sener, Urologist, Principal Investigator — Marmara University, School of Medicine, Department of Urology

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schwalb DM, Eshghi M, Davidian M, Franco I. Morphological and physiological changes in the urinary tract associated with ureteral dilation and ureteropyeloscopy: an experimental study. J Urol. 1993 Jun;149(6):1576-85. doi: 10.1016/s0022-5347(17)36456-x. PMID 8501816
- [Background] de la Rosette J, Denstedt J, Geavlete P, Keeley F, Matsuda T, Pearle M, Preminger G, Traxer O; CROES URS Study Group. The clinical research office of the endourological society ureteroscopy global study: indications, complications, and outcomes in 11,885 patients. J Endourol. 2014 Feb;28(2):131-9. doi: 10.1089/end.2013.0436. Epub 2013 Dec 17. PMID 24147820
- [Result] Sener TE, Cloutier J, Villa L, Marson F, Buttice S, Doizi S, Traxer O. Can We Provide Low Intrarenal Pressures with Good Irrigation Flow by Decreasing the Size of Ureteral Access Sheaths? J Endourol. 2016 Jan;30(1):49-55. doi: 10.1089/end.2015.0387. Epub 2015 Sep 18. PMID 26381037

RESULTS

PARTICIPANT FLOW:
Groups:
- Flexible Ureteroscopy Arm: Doppler Ultrasound examination was performed in both the pre-operative and post-operative periods on the operated kidney of patients undergoing flexible ureteroscopy + laser lithotripsy for renal stones according to EAU Guidelines
  Flexible ureteroscopy is an endourological procedure performed for kidney stones. flexible ureteroscope is a device used to reach the renal cavities through the natural urinary tract in a retrograde fashion. During operation, irrigation fluid is used to expand the cavities to provide space for movement of the device and to provide clear vision.
  Doppler Ultrasound examination: peak systolic velocities (PSV) and end diastolic velocities (EDV) of the arteries will be measured and then resistive index (RI) and pulsatility index (PI) will be calculated.
  laser lithotripsy: The laser fiber extending into the cavities through the working channel of the ureteroscope is used to fragment the stones. Laser energy is generated by the laser machine and trans
Period: Overall Study
Arm/Group | Flexible Ureteroscopy Arm
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients undergoing F-URS and laser lithotripsy for kidney stones in accordance with the EAU guidelines on Urolithiasis
Groups:
- Flexible Ureteroscopy Arm: findings of patients undergoing flexible ureteroscopy + laser lithotripsy for renal stones according to EAU Guidelines
  Flexible ureteroscopy is an endourological procedure performed for kidney stones. flexible ureteroscope is a device used to reach the renal cavities through the natural urinary tract in a retrograde fashion. During operation, irrigation fluid is used to expand the cavities to provide space for movement of the device and to provide clear vision.
  Doppler Ultrasound examination: peak systolic velocities (PSV) and end diastolic velocities (EDV) of the arteries will be measured and then resistive index (RI) and pulsatility index (PI) will be calculated.
  laser lithotripsy: The laser fiber extending into the cavities through the working channel of the ureteroscope is used to fragment the stones. Laser energy is generated by the laser machine and trans
Arm/Group | Flexible Ureteroscopy Arm
Number analyzed (Participants) | 46
Age, Continuous [Mean (Full Range); unit: years] | 41.24 [17 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 32
Body Mass Index (BMI) units: kg/m2 [Mean (Standard Deviation); unit: kg/m2] | 26.49 (4.97)
Stone volume [Mean (Full Range); unit: mm3] | 1685 [150 to 5868]

OUTCOME MEASURES:

1. Primary Outcome: Peak Systolic Velocities (PSV) Measurement by Renal Doppler Ultrasound (US) Examination Evaluating the Effects of Flexible Ureteroscopy (F-URS) on Renal Blood Flow by Demonstrating the Change Between the Pre-operative and Post-operative Parameters.
Description: Doppler US will be performed at two times: 2 days prior to surgery and within the first 24 hours following F-URS to show the change between the pre-operative and post-operative periods. Doppler examination includes renal arteries and arcuate arteries. For each patient, the following parameters are measured: peak systolic velocities (PSV) and end diastolic velocities (EDV), resistive index (RI) and pulsatility index (PI) of the arteries. The unit for PSV and EDV is cm/sec. RI and PI doesn't have a unit, they are quantitative measures calculated from PSV and EDV.
  PSV is the maximum velocity in the renal and arcuate arteries in the systolic phase of each heart pulse.
Time Frame: The doppler examination will be performed 2 days before surgery and the change will be assessed within 1 day of the operation. So, the initial evaluation will be performed and change of values will be assessed 72 hours after the initial evaluation
Measure: Median (Full Range); unit: cm/s
Groups:
- Flexible Ureteroscopy Arm: pre-operative and post-operative findings of renal Doppler Ultrasound examination on the operated kidney of patients undergoing flexible ureteroscopy + laser lithotripsy for renal stones according to EAU Guidelines
  Flexible ureteroscopy is an endourological procedure performed for kidney stones. flexible ureteroscope is a device used to reach the renal cavities through the natural urinary tract in a retrograde fashion. During operation, irrigation fluid is used to expand the cavities to provide space for movement of the device and to provide clear vision.
  Doppler Ultrasound examination: peak systolic velocities (PSV) and end diastolic velocities (EDV) of the arteries will be measured and then resistive index (RI) and pulsatility index (PI) will be calculated.
  laser lithotripsy: The laser fiber extending into the cavities through the working channel of the ureteroscope is used to fragment the stones. Laser energy is generated by the laser machine and trans
Arm/Group | Flexible Ureteroscopy Arm
Number analyzed (Participants) | 46
cm/s
  pre-operative PSV | 30.65 [18 to 82.2]
  post-operative PSV | 31.85 [16.5 to 84.1]

2. Primary Outcome: End Diastolic Velocities (EDV) Measurement by Renal Doppler Ultrasound (US) Examination Evaluating the Effects of Flexible Ureteroscopy (F-URS) on Renal Blood Flow by Demonstrating the Change Between the Pre-operative and Post-operative Parameters.
Description: Doppler US will be performed at two times: 2 days prior to surgery and within the first 24 hours following F-URS to show the change between the pre-operative and post-operative periods. Doppler examination includes renal arteries and arcuate arteries. For each patient, the following parameters are measured: peak systolic velocities (PSV) and end diastolic velocities (EDV), resistive index (RI) and pulsatility index (PI) of the arteries. The unit for PSV and EDV is cm/sec. RI and PI doesn't have a unit, they are quantitative measures calculated from PSV and EDV.
  EDV is the velocity in the renal and arcuate arteries at the end of the diastolic phase of each heart pulse.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: cm/s
Arm/Group | Flexible Ureteroscopy Arm
Number analyzed (Participants) | 46
cm/s
  pre-operative EDV | 12.3 [2.2 to 41.3]
  post-operative EDV | 12 [4.4 to 34.1]

3. Primary Outcome: Resistive Index (RI) Calculation by Renal Doppler Ultrasound (US) Examination Evaluating the Effects of Flexible Ureteroscopy (F-URS) on Renal Blood Flow by Demonstrating the Change Between the Pre-operative and Post-operative Parameters.
Description: Doppler US will be performed at two times: 2 days prior to surgery and within the first 24 hours following F-URS to show the change between the pre-operative and post-operative periods. Doppler examination includes renal arteries and arcuate arteries. For each patient, the following parameters are measured: peak systolic velocities (PSV) and end diastolic velocities (EDV), resistive index (RI) and pulsatility index (PI) of the arteries. The unit for PSV and EDV is cm/sec. RI and PI doesn't have a unit, they are quantitative measures calculated from PSV and EDV.
  Resistive index is calculated as the difference between PSV and EDV, divided by PSV [(PSV - EDV) / (PSV)].
  An increased resistive index can be considered as a marker of intrarenal arterial stiffness and is associated with worsening of renal function and tubulointersitial damage.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: unitless
Arm/Group | Flexible Ureteroscopy Arm
Number analyzed (Participants) | 46
unitless
  pre-operative RI | 0.59 [0.45 to 0.85]
  post-operative RI | 0.59 [0.41 to 0.89]

4. Primary Outcome: Pulsatility Index (PI) Calculation by Renal Doppler Ultrasound (US) Examination Evaluating the Effects of Flexible Ureteroscopy (F-URS) on Renal Blood Flow by Demonstrating the Change Between the Pre-operative and Post-operative Parameters.
Description: Doppler US will be performed at two times: 2 days prior to surgery and within the first 24 hours following F-URS to show the change between the pre-operative and post-operative periods. Doppler examination includes renal arteries and arcuate arteries. For each patient, the following parameters are measured: peak systolic velocities (PSV) and end diastolic velocities (EDV), resistive index (RI) and pulsatility index (PI) of the arteries. The unit for PSV and EDV is cm/sec. RI and PI doesn't have a unit, they are quantitative measures calculated from PSV and EDV.
  Pulsatility index is calculated as the difference between PSV and EDV, divided by the mean velocity [(PSV - EDV) / ((PSV + EDV) / 2)].
  Pulsatility index is used to discriminate between renal and pre-renal causes of acute kidney injury which can alter the therapeutic options in the clinical setting.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: unitless
Arm/Group | Flexible Ureteroscopy Arm
Number analyzed (Participants) | 46
unitless
  pre-operative PI | 0.89 [0.59 to 1.71]
  post-operative PI | 0.89 [0.54 to 1.98]

5. Secondary Outcome: Technical Details - Size of Ureteral Access Sheath
Description: The size of access sheaths will be given in French measurement. E.g. 10/12 Fr
Time Frame: 1 hour after the operation
Measure: Number; unit: participants
Groups:
- Flexible Ureteroscopy Arm: post-operative findings of renal Doppler Ultrasound examination on the operated kidney of patients undergoing flexible ureteroscopy + laser lithotripsy for renal stones according to EAU Guidelines
  Flexible ureteroscopy is an endourological procedure performed for kidney stones. flexible ureteroscope is a device used to reach the renal cavities through the natural urinary tract in a retrograde fashion. During operation, irrigation fluid is used to expand the cavities to provide space for movement of the device and to provide clear vision.
  Doppler Ultrasound examination: peak systolic velocities (PSV) and end diastolic velocities (EDV) of the arteries will be measured and then resistive index (RI) and pulsatility index (PI) will be calculated.
  laser lithotripsy: The laser fiber extending into the cavities through the working channel of the ureteroscope is used to fragment the stones. Laser energy is generated by the laser machine and trans
Arm/Group | Flexible Ureteroscopy Arm
Number analyzed (Participants) | 46
participants
  9.5/11.5 Fr | 28
  10/12 Fr | 9
  12/14 Fr | 9

6. Secondary Outcome: Technical Details - Name of Flexible Ureteroscope
Description: Each ureteroscope has unique characteristics. So, every ureteroscope that will be used, will be recorded with its name. E.g. Storz Flex-X2, Olympus V1, Wolf Cobra
Time Frame: 1 hour after the operation
Measure: Number; unit: participants
Groups:
- Flexible Ureteroscopy Arm: The type of the ureteroscope used for the flexible ureteroscopy operation
  Flexible ureteroscopy is an endourological procedure performed for kidney stones. flexible ureteroscope is a device used to reach the renal cavities through the natural urinary tract in a retrograde fashion. During operation, irrigation fluid is used to expand the cavities to provide space for movement of the device and to provide clear vision.
  Doppler Ultrasound examination: peak systolic velocities (PSV) and end diastolic velocities (EDV) of the arteries will be measured and then resistive index (RI) and pulsatility index (PI) will be calculated.
  laser lithotripsy: The laser fiber extending into the cavities through the working channel of the ureteroscope is used to fragment the stones. Laser energy is generated by the laser machine and trans
Arm/Group | Flexible Ureteroscopy Arm
Number analyzed (Participants) | 46
participants
  Storz Flex X2 | 41
  Storz Flex XC | 5

7. Secondary Outcome: Duration of the Flexible Ureteroscopy Operation
Description: the data about the duration of the operation that will be performed for each patient and the data will be recorded in minutes.
Time Frame: 10 minutes after the operation
Measure: Mean (Standard Deviation); unit: min
Groups:
- Flexible Ureteroscopy Arm: The duration of the flexible ureteroscopy operation
  Flexible ureteroscopy is an endourological procedure performed for kidney stones. flexible ureteroscope is a device used to reach the renal cavities through the natural urinary tract in a retrograde fashion. During operation, irrigation fluid is used to expand the cavities to provide space for movement of the device and to provide clear vision.
  Doppler Ultrasound examination: peak systolic velocities (PSV) and end diastolic velocities (EDV) of the arteries will be measured and then resistive index (RI) and pulsatility index (PI) will be calculated.
  laser lithotripsy: The laser fiber extending into the cavities through the working channel of the ureteroscope is used to fragment the stones. Laser energy is generated by the laser machine and trans
Arm/Group | Flexible Ureteroscopy Arm
Number analyzed (Participants) | 46
min | 62.2 (22.4)

8. Secondary Outcome: Operative Characteristics - Irrigation Pressure
Description: The pressure that is applied to the irrigation solution which is circulated through the ureteroscope that is used to expand the renal cavities during a flexible ureteroscopy operation. the data will be collected in cmH2O. This pressure value is a constant value and it doesn't change throughout the length of the procedure.
Time Frame: 1 hour after the operation
Measure: Median (Full Range); unit: cmH2O
Groups:
- Flexible Ureteroscopy Arm: The pressure applied to the irrigation solution during a flexible ureteroscopy operation
  Flexible ureteroscopy is an endourological procedure performed for kidney stones. flexible ureteroscope is a device used to reach the renal cavities through the natural urinary tract in a retrograde fashion. During operation, irrigation fluid is used to expand the cavities to provide space for movement of the device and to provide clear vision.
  Doppler Ultrasound examination: peak systolic velocities (PSV) and end diastolic velocities (EDV) of the arteries will be measured and then resistive index (RI) and pulsatility index (PI) will be calculated.
  laser lithotripsy: The laser fiber extending into the cavities through the working channel of the ureteroscope is used to fragment the stones. Laser energy is generated by the laser machine and trans
Arm/Group | Flexible Ureteroscopy Arm
Number analyzed (Participants) | 46
cmH2O | 50 [40 to 60]

9. Secondary Outcome: Operative Characteristics - Intraoperative Complications
Description: The number of patients that has experienced any kind of intraoperative complications during the flexible ureteroscopy operation.
Time Frame: 1 hour after the operation
Measure: Number; unit: participants
Groups:
- Flexible Ureteroscopy Arm: The number of patients that had a complication intraoperatively.
  Flexible ureteroscopy is an endourological procedure performed for kidney stones. flexible ureteroscope is a device used to reach the renal cavities through the natural urinary tract in a retrograde fashion. During operation, irrigation fluid is used to expand the cavities to provide space for movement of the device and to provide clear vision.
  Doppler Ultrasound examination: peak systolic velocities (PSV) and end diastolic velocities (EDV) of the arteries will be measured and then resistive index (RI) and pulsatility index (PI) will be calculated.
  laser lithotripsy: The laser fiber extending into the cavities through the working channel of the ureteroscope is used to fragment the stones. Laser energy is generated by the laser machine and trans
Arm/Group | Flexible Ureteroscopy Arm
Number analyzed (Participants) | 46
participants | 5

10. Secondary Outcome: Post-Operative Characteristics - Complications
Description: The number of patients that had a complication in the first 1 month after the operation according to the Clavien Dindo Grading system (0-5).
  Clavien Dindo Grading ranges from 0 (mildest) to 5 (most severe). 0. No complications
  1. Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Allowed therapeutic regimens are drugs as antiemetics, antipyretics, analgesics, diuretics, electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside
  2. Complications requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included
  3. Complications requiring surgical, endoscopic or radiological intervention
  4. Life-threatening complications (including CNS complications) requiring IC/ICU management
  5. Death
Time Frame: The data will be recorded within 1 month after each procedure.
Measure: Count of Participants; unit: Participants
Groups:
- Flexible Ureteroscopy Arm: The number of patients who had a complication after the flexible ureteroscopy operation in the first month following the operation.
  Flexible ureteroscopy is an endourological procedure performed for kidney stones. flexible ureteroscope is a device used to reach the renal cavities through the natural urinary tract in a retrograde fashion. During operation, irrigation fluid is used to expand the cavities to provide space for movement of the device and to provide clear vision.
  Doppler Ultrasound examination: peak systolic velocities (PSV) and end diastolic velocities (EDV) of the arteries will be measured and then resistive index (RI) and pulsatility index (PI) will be calculated.
  laser lithotripsy: The laser fiber extending into the cavities through the working channel of the ureteroscope is used to fragment the stones. Laser energy is generated by the laser machine and trans
Arm/Group | Flexible Ureteroscopy Arm
Number analyzed (Participants) | 46
Participants
  Grade 0 | 41
  Grade 1 | 3
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 1
  Grade 5 | 0

ADVERSE EVENTS:
Arm/Group | Flexible Ureteroscopy Arm
Serious Adverse Events (participants affected / at risk) | 2/46
Other Adverse Events (participants affected / at risk) | 3/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flexible Ureteroscopy Arm (N=46)
Sepsis (Renal and urinary disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flexible Ureteroscopy Arm (N=46)
Urinary tract infection (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No